CLINICAL TRIAL: NCT06528483
Title: Bladder Preservation With Sacituzumab Govitecan + Zimberelimab for Muscle-Invasive Bladder Cancer in Cisplatin-unfit and Unwilling for Cystectomy Patients: Phase II Trial
Brief Title: Bladder Preservation With Sacituzumab Govitecan + Zimberelimab for Muscle-Invasive Bladder Cancer
Acronym: preSAVE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PreSAVE INT 2024
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bladder Cancer; Bladder Urothelial Carcinoma; Bladder Neoplasm; Muscle-Invasive Bladder Carcinoma
Keywords: bladder cancer; muscle-invasive bladder cancer; bladder sparing
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — sacituzumab govitecan; zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Govitecan + Zimberelimab (Experimental): patients will be treated with Sacituzumab Govitecan 1,8q21 plus + Zimberelimab q21 for 3 cycles then radiological imaging and TURB will be repeated and patients with Stability of disease or down staging will continue Zimberelimab until disease progression, or unacceptable toxicities or completion of treatment (16 cycles). Patients with progressive disease after 3 cycles of study intervention will be treated as per clinical practice.
  Interventions: Drug: Sacituzumab Govitecan + Zimberelimab

INTERVENTIONS:
Drug: Sacituzumab Govitecan + Zimberelimab — Sacituzumab Govitecan 7.5 mg/kg IV for 3 cycles Zimberelimab 360 mg IV for 16 cycles
  Patients will be treated with Sacituzumab Govitecan 1,8q21 plus + Zimberelimab q21 for 3 cycles then radiological imaging and TURB will be repeated and patients with Stability of disease or down staging will continue Zimberelimab until disease progression, or unacceptable toxicities or completion of treatment (16 cycles). Patients with progressive disease after 3 cycles of study intervention will be treated as per clinical practice.
  Other Names: TRODELVY; AB122

SUMMARY:
Patients with MIBC N0/N1 unwilling or unfit for cystectomy will receive SG + Zimberelimab for 3 cycles of treatment prior of first radiological and TURB re-evaluation.

Patients with stable disease or downstaging will continue Zimberelimab up to 1 year. The goal of this trial is to demonstate that Sacituzumab Govitecan + Zimberelimab can avoid cistectomy and can prolong or avoid recurrence to metastatic disease in selected patients with muscle-invasive bladder cancer.

The primary endpoint of this trial is Event Free Survival that is defined as clinical evidence of new or progressing nodal or any distant metastatic disease, radical cystectomy, or death due to any cause from date of inclusion to the first documentation of a EFS event.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-group, phase 2 study. Patients with MIBC N0/N1 unwilling or unfit for cystectomy will receive SG + Zimberelimab for 3 cycles of treatment prior of first radiological and TURB re-evaluation.

Approximately 63 patients will be enrolled and assigned to study intervention. At screening, a tumor specimen from TURBT or biopsy done as early as 90 days prior to enrollment will be submitted for central pathology review. All participants will undergo baseline screening imaging (CT or MRI of the chest, abdomen, pelvis) for clinical staging.

Eligible participants will be allocated to study intervention which consist in SG + Zimberelimab for 3 cycles followed by Zimberelimab for 13 cycles in patients who achieve CR/PR/SD at tumor evaluation.

The planned total duration of treatment is approximately 1 year, 3 cycles of SG and 16 cycles of Zimberelimab.

Treatment will be discontinued if the participant experiences unacceptable AE(s), intercurrent illness that prevents further administration of treatment, the investigator's decision to withdraw the participant, the participant withdraws consent, pregnancy of the participant, noncompliance with study intervention or procedure requirements, or the maximum number of cycles has been received for each treatment component individually.

Participants will complete 3 cycles of induction study intervention, followed by repeat imaging studies (same modality as screening) within ≤4 weeks (21 days +/- 7 days) after C3D21 to exclude disease progression. mpMRI/contrast-enhanced or CT scan will assess local invasion by T3 disease or higher and the radiological response to treatment.

Participants who remain radiographically free of distant metastases and PR/SD/CR RECIST v1.1 will proceed to TURBT within 6 weeks of the last dose of SG. TURBT will enable histopathological re-staging and will evaluate pathological response to treatment. The inclusion of bladder muscle in the resection specimen is required. Cystoscopy will be performed before TURBT, as indicated in the Schedule of Activities.

Patients with no evidence of disease at the cystoscopy, will undergo bladder mapping in case of positive urine cytology. In case of negative urine cytology, patients will be considered in as complete respose, in case of no evidence of disease at radiological evaluation.

Participants with radiological progression to metastatic disease or locally advanced disease (from cT2 to cT4 or from N0 to N1), as assessed radiographically, at this time will be considered to have met the primary endpoint of EFS (ie, had an "event") and will not receive further therapy on study, but will transition into survival follow-up and will be treated as per clinical practice.

Participants with pathological downstaging and radiological complete or partial response will continue to receive zimberelimab for 13 cycles (16 cycles as a total) to complete approximately 1 year of total therapy.

Non-responder patients who will maintain radiological or pathological stability will choose to undergo RC or RT/CT or to continue Zimberelimab for 1 years. Additional TURBT could be performed in order to achieve local control, according to the centre clinical practice.

Response to study intervention will be assessed through TURBT and CT SCAN and/or MRI. Imaging should continue to be performed until an EFS event occurs or withdrawal of consent, whichever occurs first. If new anticancer therapy is initiated, this should be documented.

All subjects will be followed for OS every 3 months until death, lost to follow-up, or withdrawal of study consent. Additional survival follow-up may continue for up to 3-5 years from the time of this analysis. To evaluate metastasis free survival, subjects will be monitored by radiographic assessment and cystoscopy on an every-12-week schedule (±5 days). RECIST 1.1 criteria will be used for the assessment. Subjects will be evaluated at every SG + Zimberelimab dose administration plus two additional follow-up visits for safety within the first 100 days from the last dose of study therapy. Beyond 100 days from the last dose of study therapy, subjects will be followed for ongoing drug-related adverse events until resolved, return to baseline or deemed irreversible, or until lost to follow-up, or withdrawal of study consent.

To assess local recurrence, cystoscopy will be performed every 12 weeks (+/- 1 7 days). In case of local recurrence, patients could be managed with TURBT as per clinical practice, in case patients will still be unfit for cystectomy or refuse surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years old of age, at the time of providing informed consent.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Patients deemed ineligible for Radical Cystectomy (RC) + Retroperitoneal lymphnode dissection (RPNLD) by a urologist and/or oncologist and/or anesthesiology.
* Cisplatin unfit patients as per Galsky criteria (ECOG Performance Status of 2 and/or creatinine-clearance < 60 ml/min and/or CTCAE Gr ≥ 2 hearing loss and/or CTCAE Gr ≥ 2 neuropathy).
* Cisplatin-fit patients are admitted if they are unwilling to undergo Radical Cystectomy (RC) and unwilling for cisplatin-based chemotherapy.
* Patients deemed eligible for surgery will be included if they will be unwilling to undergo RC and will be ineligible and/or unwilling to cisplatin-based chemotherapy.
* cT2-cT4 bladder cancer patients with predominant urothelial histology or Squamous cell histologic variant with histological confirmed diagnosis of muscle-invasive bladder cancer (MIBC) obtained via a diagnostic or maximal TURBT performed within 90 days before enrollment.
* cN0-1 bladder cancer patients with predominant urothelial histology or Squamous cell histologic variant
* Have adequate organ function as defined as follow (Specimens must be collected within 10 days prior to the start of study intervention):

  * Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study treatment initiations (hemoglobin ≥ 9 g/dL, ANC ≥ 1500/mm3, and platelets ≥ 100,000/μL).
  * Adequate hepatic function (bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5 × ULN or ≤ 5 × ULN if known liver metastases, and serum albumin > 3 g/dL).
  * Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation.
  * International normalized ratio (INR)/PT and PTT or aPTT ≤ 1.5 ULN unless patient is currently receiving therapeutic anticoagulant therapy.
* Patients with HIV must be on antiretroviral therapy (ART) and have a well-controlled

HIV infection/disease defined as:

* Patients on ART must have a CD4+ T-cell count ≥ 350 cells/mm3 at time of screening.
* Patients on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening.
* Patients on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).
* The combination ART regimen must not contain any medications that may interfere with SN-38 metabolism.

Exclusion Criteria:

1. Positive serum pregnancy test (Appendices 9.4) or women who are breastfeeding.
2. Known hypersensitivity to the study drug, its metabolites, or formulation excipient.
3. Requirement for ongoing therapy with or prior use of any prohibited medications listed in Section.
4. Have had a prior anticancer biologic agent within 4 weeks prior to enrollment or have had prior chemotherapy or targeted small molecule therapy. Patients participating in observational studies are eligible.
5. Have previously received topoisomerase 1 inhibitors.
6. Have an active second malignancy. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll. Other exception are localized prostate cancer with a Gleason score of 6 (treated within the last 24 months or untreated and under surveillance) and localized prostate cancer with a Gleason score of 3+4 that has been treated more than 6 months prior to full study screening and considered to have a very low risk of recurrence.
7. Patients with neuroendocrine histology will be excluded.
8. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
9. Have active serious infection requiring antibiotics.
10. Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
11. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

    * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
    * Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
12. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
13. Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study.
14. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | 24 months
  clinical evidence of new or progressing nodal or any distant metastatic disease, radical cystectomy, or death due to any cause from date of inclusion to the first documentation of a EFS event. Patients last known to be EFS event-free are censored at the date of last event-free cystoscopy and/or CT scan. Those patients without disease assessment who are still alive will be censored at date of inclusion in the trial

SECONDARY OUTCOMES:
clinical or pathological downstaging | 24 months
  Participants experiencing partial response according to RECIST v1.1 criteria and/or pathological downstaging as from pT2 to non muscle-invasive disease after SG + Zimberelimab treatment
Number of Participants treated with Pembrolizumab + Enfortumab Vedotin who experience AEs/SAEs | 24 months
  The incidence of, causality, and outcome of AEs/SAEs. AEs will be assessed as defined by CTCAE, Version [5.0]
predictive role of miRNA in patients who achieve clinical or pathological downstaging after SG + Zimberelimab treatment | 24 months
  miRNA expression in partecipants who achieve clinical or pathological downstaging after SG + Zimberelimab treatment
predictive role of ctDNA in patients who achieve clinical or pathological downstaging after SG + Zimberelimab treatment | 24 months
  • ctDNA expression in partecipants who achieve clinical or pathological downstaging after SG + Zimberelimab treatment
role of 18FDG-PET in the prediction of response or relapse for N positive patients | 24 months
  Patients experiencing nodal progression or remission after SG + ZIM treatment
the role of multiparametric MRI (mpMRI) in the assessment of clinical response | 24 months
  Patients with tumor response identified by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione Irccs Istituto Nazionale Dei Tumori Di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bokarica P, Hrkac A, Gilja I. Re: J. Alfred Witjes, Thierry Lebret, Eva M. Comperat, et al. Updated 2016 EAU Guidelines on Muscle-invasive and Metastatic Bladder Cancer. Eur Urol 2017;71:462-75. Eur Urol. 2017 Aug;72(2):e45. doi: 10.1016/j.eururo.2017.02.031. Epub 2017 Mar 6. No abstract available. PMID 28279514
- [Background] Softness K, Kaul S, Fleishman A, Efstathiou J, Bellmunt J, Kim SP, Korets R, Chang P, Wagner A, Olumi AF, Gershman B. Radical cystectomy versus trimodality therapy for muscle-invasive urothelial carcinoma of the bladder. Urol Oncol. 2022 Jun;40(6):272.e1-272.e9. doi: 10.1016/j.urolonc.2021.12.015. Epub 2022 Jan 17. PMID 35058142
- [Background] Royce TJ, Feldman AS, Mossanen M, Yang JC, Shipley WU, Pandharipande PV, Efstathiou JA. Comparative Effectiveness of Bladder-preserving Tri-modality Therapy Versus Radical Cystectomy for Muscle-invasive Bladder Cancer. Clin Genitourin Cancer. 2019 Feb;17(1):23-31.e3. doi: 10.1016/j.clgc.2018.09.023. Epub 2018 Oct 4. PMID 30482661
- [Background] Mitin T, Hunt D, Shipley WU, Kaufman DS, Uzzo R, Wu CL, Buyyounouski MK, Sandler H, Zietman AL. Transurethral surgery and twice-daily radiation plus paclitaxel-cisplatin or fluorouracil-cisplatin with selective bladder preservation and adjuvant chemotherapy for patients with muscle invasive bladder cancer (RTOG 0233): a randomised multicentre phase 2 trial. Lancet Oncol. 2013 Aug;14(9):863-72. doi: 10.1016/S1470-2045(13)70255-9. Epub 2013 Jul 1. PMID 23823157
- [Background] James ND, Hussain SA, Hall E, Jenkins P, Tremlett J, Rawlings C, Crundwell M, Sizer B, Sreenivasan T, Hendron C, Lewis R, Waters R, Huddart RA; BC2001 Investigators. Radiotherapy with or without chemotherapy in muscle-invasive bladder cancer. N Engl J Med. 2012 Apr 19;366(16):1477-88. doi: 10.1056/NEJMoa1106106. PMID 22512481
- [Background] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte R, Wang J, Huang B, Davis C, Fowst C, Costa N, Blake-Haskins JA, di Pietro A, Grivas P. Avelumab Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2020 Sep 24;383(13):1218-1230. doi: 10.1056/NEJMoa2002788. Epub 2020 Sep 18. PMID 32945632
- [Background] Powles T, Bellmunt J, Comperat E, De Santis M, Huddart R, Loriot Y, Necchi A, Valderrama BP, Ravaud A, Shariat SF, Szabados B, van der Heijden MS, Gillessen S; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Bladder cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2022 Mar;33(3):244-258. doi: 10.1016/j.annonc.2021.11.012. Epub 2021 Nov 30. No abstract available. PMID 34861372
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Lin N, Zhang M, Bai H, Liu H, Cui J, Ke X, Zhang H, Liu L, Yan D, Jiang Y, Zang A, Qi J, Wang L, Liu Z, Xu B, Zhang Y, Zhang Z, Zhao X, Hu C, Yang S, Zhou H, Shi J, Shao Z, Xiang Y, Zhu J, Song Y, Zhu J. Efficacy and safety of GLS-010 (zimberelimab) in patients with relapsed or refractory classical Hodgkin lymphoma: A multicenter, single-arm, phase II study. Eur J Cancer. 2022 Mar;164:117-126. doi: 10.1016/j.ejca.2021.07.021. Epub 2021 Aug 27. PMID 34462189
- [Background] Loriot Y, Petrylak DP, Rezazadeh Kalebasty A, Flechon A, Jain RK, Gupta S, Bupathi M, Beuzeboc P, Palmbos P, Balar AV, Kyriakopoulos CE, Pouessel D, Sternberg CN, Tonelli J, Sierecki M, Zhou H, Grivas P, Barthelemy P, Tagawa ST. TROPHY-U-01, a phase II open-label study of sacituzumab govitecan in patients with metastatic urothelial carcinoma progressing after platinum-based chemotherapy and checkpoint inhibitors: updated safety and efficacy outcomes. Ann Oncol. 2024 Apr;35(4):392-401. doi: 10.1016/j.annonc.2024.01.002. Epub 2024 Jan 18. PMID 38244927
- [Background] Grivas P, Pouessel D, Park CH, Barthelemy P, Bupathi M, Petrylak DP, Agarwal N, Gupta S, Flechon A, Ramamurthy C, Davis NB, Recio-Boiles A, Sternberg CN, Bhatia A, Pichardo C, Sierecki M, Tonelli J, Zhou H, Tagawa ST, Loriot Y. Sacituzumab Govitecan in Combination With Pembrolizumab for Patients With Metastatic Urothelial Cancer That Progressed After Platinum-Based Chemotherapy: TROPHY-U-01 Cohort 3. J Clin Oncol. 2024 Apr 20;42(12):1415-1425. doi: 10.1200/JCO.22.02835. Epub 2024 Jan 23. PMID 38261969